# **Statistical Analysis Plan (SAP)**

# Development of a Normative Database for Rheumatoid Arthritis (RA) Imaging with Tc 99m Tilmanocept

Study No: NAV3-35

Version 1.0

July 14, 2022

Prepared for Navidea Biopharmaceuticals, Inc. 4995 Bradenton Avenue, Suite 240 Dublin, OH 43017

Prepared by STATKING Clinical Services 759 Wessel Drive Fairfield, OH 45014 513-858-2989 www.statkingclinical.com



# **Approval Page**

By entering into this Statistical Analysis Plan (SAP), the parties acknowledge and agree that this SAP shall be incorporated into and subject to the terms of the Master Services Agreement (MSA). Any changes requested by Client to this SAP shall be subject to Section I.C of the MSA requiring a mutually agreed upon "Change Order" prior to any modification of the procedures set forth herein.

I agree to the format and content of this document.

| Approved by: | |
|------------------------------------------|--------------|
| Michael Rosol, PhD Chief Medical Officer | 20 July 2022 |
| Navidea Biopharmaceuticals | |
| 4995 Bradenton Avenue, Suite 240 | |
| Dublin, Ohio 43017 | |
| MRosol@navidea.com | |

20 July 2022 Date Rachael Surshan Rachael Hershey, MS, CCRP

Associate Director, Clinical Research & Operations Navidea Biopharmaceuticals 4995 Bradenton Avenue, Suite 240 Dublin, Ohio 43017

RHershey@navidea.com

Authored by:

lan Lees, MS Statistician

STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 327 ian@statkingclinical.com

07/21/2022

Approved by (internal review):

Lori Christman, PhD
Director of Biostatistics
STATKING Clinical Services

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 330 lori@statkingclinical.com Date 21 2022

7-20-2022

Approved by:

Clare Geiger, RN Project Manager

**STATKING Clinical Services** 

759 Wessel Drive Fairfield, OH 45014 513-858-2989 ext. 304 clare@statkingclinical.com Date

# **Revision History**

Not Applicable.

# **List of Abbreviations and Definitions of Terms**

| Term | Definition |
|---|---|
| Δ | Greek letter delta, used to represent the change in a |
| | particular variable |
| μg | microgram |
| ACPA | anti-citrullinated protein/peptide antibody |
| ACR/EULAR | American College of Rheumatology/ European League |
| | Against Rheumatism |
| AE | adverse event |
| Anti-TNF-α | Anti-Tumor Necrosis Factor $\alpha$ biological Disease Modifying |
| bDMARD | Anti-Rheumatic Drug |
| CDAI | Clinical Disease Activity Index |
| CFB | change from baseline |
| CI | confidence interval |
| CRF | case report form |
| CSR | clinical study report |
| CT | X-ray computed tomography |
| CV | coefficient of variation |
| DAS28 | Disease activity score used with the ACR/EULAR 2010 RA |
| | guidelines |
| ECG | electrocardiogram |
| FDA | Food and Drug Administration |
| HAQ-DI | Health Assessment Questionnaire Disability Index |
| HC(s) | healthy control(s) |
| ICH | International Conference on Harmonization |
| ITD | intent-to-diagnose |
| IV | intravenous |
| mCi | milliCurie (37x10 <sup>6</sup> becquerels; 37megabecquerels) |
| MCP | metacarpophalange |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NPV | Negative Predictive Value |
| OA | Osteoarthritis or Overall Accuracy, depending on context |
| PIP | proximal interphalange |
| PP | per protocol |
| PPV | Positive Predictive Value |
| RA | rheumatoid arthritis |
| ROI | region of interest |
| RR | reference region |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | system organ class |
| SPECT | single photon emission computed tomography |

| Term | Definition |
|---|---|
| Tc 99m | technetium-99m metastable isotope; γ-emitting (half-life |
| | 6.02 h) |
| TEAE | treatment-emergent adverse event |
| TESAE | treatment-emergent serious adverse event |
| tilmanocept | DTPA Mannosyl Dextran (the US Adopted Name for the |
| | drug substance of Lymphoseek) |
| TUV | Tilmanocept uptake value |
| US | United States |
| $\bar{X}_{BRAIN}$ | the decay-corrected average voxel intensity of the brain |
| | RR of a subject at the anterior view at 1 or 3-hours post- |
| | injection |
| $\bar{X}_{ROI}$ | the decay-corrected average voxel intensity of a region of |
| | interest |

# **Table of Contents**

| APPROVAL PAGE | 1 |
|------------------------------------------------------|----|
| REVISION HISTORY | 4 |
| LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 5 |
| INTRODUCTION | 9 |
| 1.0 SYNOPSIS OF STUDY DESIGN/PROCEDURES | 9 |
| 1.1 Design and Treatment | 10 |
| 1.2 Study Procedures | 10 |
| 1.3 Sample Size | 11 |
| 2.0 DATA ANALYSIS CONSIDERATIONS | 12 |
| 2.1 Types of Analyses | 12 |
| 2.2 Analysis Populations | 12 |
| 2.3 Missing Data Conventions | 13 |
| 2.4 Interim Analyses | 13 |
| 2.5 Calculation of TUV | 13 |
| 2.6 Study Center Considerations in the Data Analysis | 14 |
| 2.7 Documentation and Other Considerations | 14 |
| 3.0 ANALYSIS OF BASELINE PATIENT CHARACTERISTICS | 15 |
| 4.0 ANALYSIS OF EFFICACY | 15 |
| 4.1 Description of Efficacy Endpoints | 15 |
| 4.2 Analysis of Efficacy Variables | 17 |
| 5.0 ANALYSIS OF SAFETY | 18 |
| 5.1 Description of Safety Variables | 18 |

| 5.2 Description of Safety Analysis | 18 |
|---------------------------------------------------------|----|
| 6.0 OTHER RELEVANT DATA ANALYSES/SUMMARIES | 20 |
| 6.1 Patient Completion | 20 |
| 6.3 Study Drug Administration | 20 |
| 6.4 RA Evaluation | 20 |
| 6.5 Concomitant Medications | 20 |
| 7.0 LIST OF ANALYSIS TABLES, FIGURES AND LISTINGS | 21 |
| 8.0 REFERENCES | 25 |
| APPENDIX A – TABLES, FIGURES AND LISTING SPECIFICATIONS | 26 |
| APPENDIX B – TABI F SHFI I S | 28 |

#### INTRODUCTION

#### **Description**

This Statistical Analysis Plan (SAP) is consistent with the final study protocol (dated 17 March 2021) and includes the latest details of efficacy and safety summaries to be included in the clinical study report (CSR).

The preparation of this SAP was done in accordance with STATKING Clinical Services SOP SCI 02-54, Statistical Analysis Plans.

# 1.0 Synopsis of Study Design/Procedures

This is a prospective, open-label, multicenter, single-dose study designed to develop a normative database of joint-specific Tilmanocept Uptake Values ( $TUV_{joint}$ ) in healthy controls (HCs) and to assess the feasibility of qualitative and quantitative single photon emission computed tomography/ computed tomography (SPECT/CT) assessments in HCs and subjects with active rheumatoid arthritis RA following Tc 99m tilmanocept administration.

Tilmanocept Uptake Value (TUV) is a quantitative imaging metric used to characterize Tc 99m tilmanocept uptake on planar imaging. A per-joint TUV (TUV $_{\rm joint}$ ) relative ratio will be calculated for the each of the 22 DAS28 joints located in the hands and wrists. A subject-level global TUV (TUV $_{\rm global}$ ) assessed across the 22 joints will be used as an indication of overall disease burden in RA patients.

The study is stratified into two arms. Arm 1 consists of HC subjects. Arm 2 consists of HCs and clinically diagnosed RA patients on stable therapy.

The objectives of the study are:

#### **Primary Objectives:**

- To establish mean and variance of TUV<sub>joint</sub> in HCs age-matched to RA population.
- To assess the feasibility of detecting Tc 99m tilmanocept anatomic localization using SPECT/CT imaging of hands and wrists in HCs and subjects with active RA.

#### Secondary Objectives:

• To quantitate Tc 99m tilmanocept anatomic localization based on SPECT/CT imaging of hands and wrists in HCs and joints with RAinvolved inflammation.

## Safety Objective:

 To evaluate safety through the examination of adverse event (AE) incidence and changes over time in laboratory tests, vital signs, and physical examination findings.

#### 1.1 Design and Treatment

Subjects will receive the administration of Tc 99m tilmanocept through an IV route of administration. All subjects will receive a 150 µg mass dose of tilmanocept labeled with 10 mCi of Tc 99m in a 3 ml volume. Following injection a 10 ml sterile normal saline flush will be administered. The preferred site of IV placement will be the left or right antecubital vein.

| Tabl | le 1 | Study | arms |
|------|------|-------|------|
|------|------|-------|------|

| Table 1 Study | y arms | |
|---|---|---|
| Arm | Subjects | Evaluations |
| 1 | HC subjects clinically free of any inflammatory disease and/or joint pain. | Planar image of bilateral hands/wrists. |
| 2 | HC subjects clinically free of any inflammatory disease and/or joint pain. Subjects with clinically diagnosed RA who have been on stable anti-rheumatic therapy. | Planar image of<br>bilateral<br>hands/wrists followed<br>by SPECT/CT of<br>bilateral hands/wrists. |

### 1.2 Study Procedures

Subjects will visit the study site (Visit 1) for screening procedures up to 30 days (Day -30 to Day -1) before enrollment into the study. Screening procedures (demographics, vital signs, medical history, blood and urine samples for clinical labs, RA specific labs, urine pregnancy testing for subjects of childbearing potential, and physical exam) will be completed along with the 2010 ACR/EULAR score. RA subjects will also undergo a DAS28 evaluation and a review of RA history including previous treatments, date of symptom onset, and date of diagnosis.

Subjects arriving for Study Day 0 (Visit 2) will be considered enrolled in the study. On Day 0 subjects will receive Tc 99m injection and imaging procedures. A urine pregnancy test will be administered (pre-injection) to all subjects with childbearing potential. Up to 30 minutes prior to drug administration assessment of vital signs and AEs will be performed. After pre-injection procedures are completed subjects will receive a single IV dose with 150  $\mu g$  of tilmanocept radiolabeled with 10 mCi of Tc 99m. Within 30 minutes of injection, subjects will receive vital sign and AE check. For all subjects, planar images of the bilateral hands and wrists will be taken at 60 - 75 minutes for 10 – 13 minutes. After preparation up to 10 minutes, for Arm 2, SPECT/CT of the bilateral hands and wrists will be acquired for 25-30 minutes.

On Study Day 5 ( $\pm$  3 days) (Visit 3) a safety follow-up telephone call will include a review of concomitant medications and assessment of adverse events. Subjects have completed the study at this point.

For all subjects, delegated trained imaging scientists blinded to all clinical subject information will perform semi-automated region-of-interest ROI drawing on planar images of the bilateral hands and wrists to derive relevant count statistics, which are input parameters for TUV<sub>joint</sub> and TUV<sub>global</sub>.

#### 1.3 Sample Size

The study will enroll up to 135 evaluable subjects in Arms 1 and 2 allocated below, imaged at up to 8 study centers.

Arm 1 will have up to N = 120 evaluable HC subjects, Arm 2 will have up to N = 15 evaluable subjects; 5 HCs and 10 RA subjects.

A subject is considered evaluable if he/she meets the criteria for the analysis population and has the data necessary for computing the primary endpoint(s) relevant to his/her study Arm.

The sample will be stratified 3:1, females to males ratio to reflect RA incidence in the United States. The sex-specific samples will be further stratified by age to reflect the Census estimated US population in 2019.

The target sample sizes are given below.

| Age Range | Male | Female | Total |
|--------------------|------|--------|-------|
| 30 to 39 years | 8 | 23 | 31 |
| 40 to 49 years | 7 | 21 | 28 |
| 50 to 59 years | 8 | 22 | 30 |
| 60 to 69 years | 7 | 21 | 28 |
| 70 years and older | 6 | 21 | 27 |
| Total | 36 | 108 | 144 |

An effort will be made to target enrollment in this group to include 2 men and 8 women 80 years old and over.

The existing data for HC subjects was used in a bootstrap procedure to evaluate the width of 95% confidence intervals for the 95 percentiles for various sample sizes. The sponsor has decided for its business purposes that knowing the percentile to within 0.05 of its true value is sufficient. A sample of size N = 144 HC results (this includes the subjects from Arm 1 of NAV3-31) in 95% confidence intervals with half-widths less than 0.05.

The sample size for Arm 2 was determined to be sufficient for the business purposes of the sponsor. The sample size for Arm 2 will be 5 HCs and 10 RA subjects.

# 2.0 Data Analysis Considerations

#### 2.1 Types of Analyses

Data analyses described in this SAP will consist of analyzing efficacy and safety data.

#### 2.2 Analysis Populations

The following analysis populations will be used in the study:

**Safety Population** – The safety population includes all patients that have been enrolled in the study and injected with Tc 99m tilmanocept.

**Intent-to-Diagnose (ITD) Population** – The ITD population includes all subjects that have been enrolled in the study, injected with Tc 99m tilmanocept, and

received all imaging and evaluations necessary for the primary endpoint(s) appropriate to their respective arm.

**Per Protocol (PP) Population:** The PP population will include all ITD subjects without major protocol violations. All protocol violations will be classified as major or minor prior to database lock.

All efficacy analyses will be carried out on the ITD and PP populations with the ITD population being the primary analysis set. All analyses of safety data and baseline subject characteristics will be carried out on the safety population. A data listing displaying the patients excluded from each population will be created, as shown in Appendix B.

#### 2.3 Missing Data Conventions

No missing value imputation will be used in this analysis. All analyses will be based on the observed data.

#### 2.4 Interim Analyses

There are no interim analyses planned for this study.

#### 2.5 Calculation of TUV

All calculations are done on a reader-specific basis. That is, there is no statistical aggregation of the reader results.

#### Calculating Joint TUV

For an individual joint,  $TUV_{joint}$  is defined as the average pixel intensity of the joint (ROI) divided by the average pixel intensity of the whole hand and part of the forearm on the same view and side as the joint ROI.

#### **Calculating Global TUV**

For each independent blind reader, determine the average  $TUV_{joint}$  and 95% prediction interval of both the anterior and posterior views of the wrists, MCPs, and PIPs in healthy individuals. For all following calculations, reader specific average  $TUV_{joint}$  and 95% prediction intervals will be used.

For each RA subject do the following.

Step 1: Calculate TUV<sub>joint</sub> for each of the 22 DAS28 joints for which data are collected.

Step 2: Identify all imaged joints with  $TUV_{joint}$  > upper limit of normal for the anatomically similar joint and view. These will be referred to as inflamed joints (IJ). Each joint has an anterior and posterior view: a joint is considered an IJ if either view has a  $TUV_{joint}$  higher than the upper bound from the normative data set.

Step 3: Calculate the macrophage-involved contribution (MI) to Tc 99m tilmanocept localization for each IJ. This is done by expressing the TUV for the IJ as a fractional change from the mean TUV for the anatomically equivalent joint and view. That is, if  $TUV_{joint}$  and  $\overline{H}_{joint}$  represent the joint and view specific TUV and the mean TUV for the anatomically equivalent joint and view from the normative data set respectively, the macrophage contribution to TUV is  $Ml_{joint}$ :

$$MI_{joint} = \frac{TUV_{joint} - \overline{H}_{joint}}{\overline{H}_{joint}}.$$

Step 4:  $TUV_{global}$  is the total of the macrophage-involved contributions for the IJs. (Note that  $MI_k$  is effectively 0 if  $TUV_{joint}$  is less than or equal to the upper limit of normal from the normative data set.) That is,

$$TUV_{global} = \sum_{All IIs} MI_{IJ} = \sum_{k=1}^{22} MI_k.$$

Arms 1 and 2:

Precision endpoints for both arms will be assessed estimating the mean, standard deviation, n, minimum, median, and maximum of TUV for each evaluated DAS28 joint.

#### 2.6 Study Center Considerations in the Data Analysis

A study center is defined as a treatment administration site or group of treatment administration sites under the control and supervision of the same Principal Investigator (PI). There will be no selective pooling of study centers.

#### 2.7 Documentation and Other Considerations

The data analyses described in this SAP will be conducted using SAS<sup>©</sup> Software, version 9.4 or later.

# 3.0 Analysis of Baseline Patient Characteristics

Baseline and demographic characteristics of the safety population will be summarized by subject arm and overall. Continuous variables (age, height, and weight) will be summarized via mean, standard deviation, minimum, maximum, and number of non-missing responses. Categorical variables (gender, race, and ethnicity) will be summarized via counts and percentages.

A detailed listing of baseline data for each patient in the safety population will also be provided, as shown in Appendix B.

# 4.0 Analysis of Efficacy

### 4.1 Description of Efficacy Endpoints

The efficacy variables for this study are as follows:

- Quantitative determination of TUV<sub>joint</sub> and TUV<sub>global</sub>.
- Qualitative determination of tilmanocept localization in planar images and SPECT/CT images of the bilateral hands and wrists.
- Quantitative determination of tilmanocept localization in planar and SPECT/ CT images of the bilateral hands and wrists

The presence of radiotracer uptake for a joint indicates the presumed presence of activated macrophages. The use of the term "localization" in this SAP is synonymous with the presence of radiotracer uptake.

TUV is defined as:

$$TUV_{joint} = \frac{\bar{X}_{joint}}{\bar{X}_{RR}};$$

where

- $\bar{X}_{joint}$  is the average voxel intensity of a particular joint of a subject at the anterior or posterior views at 1 hour post-injection.
- $\bar{X}_{RR}$  is the average voxel intensity of the reference region (RR) of a subject at the anterior or posterior views at 1 hour post-injection.

# 4.1.1 Primary Efficacy Endpoints

The primary efficacy endpoints of this study are:

#### Arm 1:

The normal limits of TUV<sub>joint</sub> per joint basis in HC subjects, which are defined as the 5 and 95 percentiles of TUV<sub>joint</sub> of bilateral joints (i.e., bilateral wrists, metacarpophalangeal joint [MCPs], proximal interphalangeal [PIPs]). The normal range will be determined separately for each of the three blinded readers.

#### Arm 2:

The qualitative evaluations of planar and SPECT/CT in detecting localization within synovial spaces of the bilateral hands and wrists in HCs and RA subjects.

### 4.1.2 Secondary efficacy Endpoints

The Secondary efficacy endpoints of this study are:

Healthy Controls in Both Arms 1 and 2:

- Applicability of the Normal (Gaussian) distribution to TUV<sub>joint</sub> data.
- Relationship between TUV<sub>joint</sub> and age by joint.
- Relationship between the variance of TUV<sub>joint</sub> and age.
- Relationship between TUV<sub>joint</sub> and sex (male vs female).
- Relationship between TUV<sub>joint</sub> and BMI.

#### Arm 2:

- Quantitative evaluations of Tc 99m tilmanocept localization from SPECT/CT within synovial spaces of the bilateral hands and wrists in HCs and RA subjects.
- Normative joint-specific standardized uptake value (SUV).
- Predictive value of planar scans for SPECT/CT scans.

#### 4.2 Analysis of Efficacy Variables

#### 4.2.1 Analysis of Primary Efficacy Variables

#### Arm 1:

All TUV<sub>joint</sub> data will be analyzed with summary statistics (mean, standard deviation, n, minimum, median, maximum) by reader, joint and view.

The 5 and 95 percentiles will be estimated with quantile regression fitting an intercept as a fixed term. The lower and upper limits of normal TUV<sub>joint</sub> will be determined using non-parametric confidence intervals and kernel density-based confidence intervals.

#### Arm 2.

Localization of tilmanocept in the hands and wrists will be summarized with frequency counts and percentages by reader and joint.

#### 4.2.2 Analysis of Secondary Efficacy Variables

Healthy Controls in Both Arms 1 and 2:

Normal quantile plots will be provided per-joint and reader, along with the p-value for the Shapiro-Wilk test of Normality.

Scatter plots of  $TUV_{joint}$  by age per-joint will be provided, along with the correlation coefficients and p-values. The hypotheses for the p-value to test the correlation coefficient are:  $H_0$ :  $\rho = 0$  vs  $H_1$ :  $\rho \neq 0$ , where  $\rho$  is the correlation coefficient. The p-value evaluating age in the regression model will be provided in the figure.

Scatter plots of  $TUV_{joint}$  by BMI will be provided, along with the correlation coefficients and p-values. The hypotheses for the p-value to test the correlation coefficient are:  $H_0$ :  $\rho = 0$  vs  $H_1$ :  $\rho \neq 0$ , where  $\rho$  is the correlation coefficient. The p-value evaluating BMI in the regression model will be provided in the figure.

Scatter plots of TUV<sub>joint</sub> by sex will be provided.

To check the relationship between the variance of TUV<sub>joint</sub> and age, a quantile regression model will be fitted with an intercept as a fixed term. The plot of the residuals on the y-axis and age on the x-axis will be provided.

#### Arm 2:

SUV will be calculated and summarized on both a per-joint and a total of all joints with summary statistics: mean, standard deviation, n, minimum, maximum, and median. The formula for SUV is:

$$SUV = \frac{r}{(a'/w)};$$

where:

r: The radioactivity activity concentration [kBq/mL]

a': The decay-corrected amount of injected radiolabeled FDG [kBq]

w: The weight of the patient [g]

The predictive value of planar scans for SPECT/CT qualitative findings will be summarized per joint and reader with a crosstabulation and the uncertainty coefficients for row | column, column | row, and symmetric. The planar result will be deemed "positive" (i.e., inflamed) if TUV<sub>joint</sub> > 95 percentile of the reader.

# 5.0 Analysis of Safety

#### 5.1 Description of Safety Variables

The safety analysis variables are defined as follows:

- Adverse Events (AEs)
- Clinical Laboratory Tests (hematology, serum chemistry, urinalysis, RA panel)
- Vital Signs

#### 5.2 Description of Safety Analysis

The following describes the safety analyses to be performed for the study. All safety analyses will be performed on the safety population. Follow up timing will vary by arm as noted above.

#### **Adverse Events**

Adverse events will be observed for each subject from signing of informed consent until termination from the study. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®). A treatment-emergent AE (TEAE) is defined as an AE whose start date is on or after the initial procedure date. Based on the coded terms, frequencies of each TEAE will be summarized by MedDRA® preferred term within system organ class (SOC), by severity grade, and by relationship to Tc 99m Tilmanocept for each arm and overall.

A summary of TEAEs will be constructed showing the following by arm and overall:

- Number of subjects with at least one TEAE
- TEAEs by arm and severity grade
- TEAE by arm and relationship to Tc 99m tilmanocept
- TEAEs by arm and relationship of TEAE to study procedure
- Number of subjects with at least one treatment emergent serious adverse event

Treatment-emergent serious adverse events (TESAEs) will be tabulated by MedDRA® preferred term within SOC by arm and overall.

A by-patient AE data listing of all AEs including verbatim term, coded term, grade, and relation to study drug will be provided.

## **Clinical Laboratory Tests**

Clinical laboratory tests will be performed at screening (baseline) and after the final image acquisition on the imaging day. Only abnormal laboratory values and RA lab values will be assessed for clinical significance as applicable. For each quantitative laboratory test, summary statistics (mean, standard deviation, median, range, n) on the raw as well as their changes from baseline will be presented by timepoint, by arm, and overall. A shift table will also be produced to show the changes in lab values over time relative to the normal ranges.

If multiple labs were performed at a given visit, then the latest results will be summarized in the analysis tables. All collected lab data will be listed.

#### **Vital Signs**

Vital signs will be performed at screening, just prior to and just after injection. Height and weight will be measured only at screening and will be summarized as part of the baseline and demographic information. For each vital sign (respiration rate, systolic blood pressure, diastolic blood pressure, heart rate and temperature), summary statistics (mean, standard deviation, minimum, maximum, n) on the raw as well as their changes from baseline will be presented by timepoint, by arm, and overall. The baseline value for each of the post-injection vital sign parameters will be the corresponding pre-injection time point. If there are multiple vital signs taken at any time point, then the latest set of vital signs will be used for the analysis. All vital sign data will be listed.

# 6.0 Other Relevant Data Analyses/Summaries

# **6.1 Patient Completion**

A table will be constructed with counts of screen failures and enrolled subjects. Of those enrolled, counts and percentages of patients withdrawing from the study before study completion and the number completing the study will be displayed. For those subjects that withdraw before completion of the study, counts and percentages of the reasons for withdrawal will be tabulated. The table will include summary counts and percentages by study arm and overall. A data listing of all subject completion and withdrawal data will also be constructed.

#### 6.2 Physical Exam

Physical exams will be performed at screening. All physical exam data will be listed.

#### **6.3 Study Drug Administration**

The volume, the calculated mass dose, and radioactivity of Tc 99m tilmanocept injected will be summarized by arm and overall. All study drug administration data will be listed.

#### 6.4 RA Evaluation

Each RA subject will undergo a DAS28 evaluation during screening. The swollen and tender joints will be identified and documented during the physical examination. Results of all DAS28 evaluations will be listed.

#### 6.5 Concomitant Medications

Prior and concomitant medications will be collected for 30 days prior to Day 0, and all RA medications will be collected for 6 months prior to Day 0. All prior and concomitant medications will be listed, as shown in Appendix B. A separate data listing will be created to show only those medications that were taken for RA within the 6 months prior to Day 0 injection.

# 7.0 List of Analysis Tables, Figures and Listings

| Table<br>No. | Table Title | Included in Final Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 1 | Subject Disposition by Study Arm | X | X |
| 2 | Demographics and Baseline Data Summary Statistics by Arm – Continuous Variables (Safety Population) | Х | Х |
| 3 | Demographics and Baseline Data Summary Statistics by Arm – Categorical Variables (Safety Population) | Х | Х |
| 4 | Summary of Study Drug Administration by Arm (Safety Population) | Х | Х |
| 5 | Summary of TUV <sub>joint</sub> on both Arms Per Reader, Joint, and View (ITD population) | Х | Х |
| 6 | Summary of TUV <sub>joint</sub> on both Arms Per Reader, Joint, and View (PP Population) | Х | |
| 7 | Summary of SUV on Arm 2 per Joint and a Total of All Joints (ITD population) | Х | Х |
| 8 | Summary of SUV on Arm 2 per Joint and a Total of All Joints (PP Population) | Х | |
| 9 | Normal Range of TUV <sub>joint</sub> for the Three Blinded Readers in All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | Х |
| 10 | Normal Range of TUV <sub>joint</sub> for the Three Blinded Readers in All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| 11 | Correlation Between TUV <sub>joint</sub> and Age and BMI – All Arm 1 and 2<br>Healthy Control Subjects (ITD Population) | Х | Х |
| 12 | Correlation Between TUV <sub>joint</sub> and Age and BMI – All Arm 1 and 2<br>Healthy Control Subjects (PP Population) | Х | |
| 13 | Frequency Counts and Percentage of Localization in SPECT/ CT Imaging in RA Subjects (ITD Population) | Х | Х |
| 14 | Frequency Counts and Percentage of Localization in SPECT/ CT Imaging in RA Subjects (PP Population) | X | |
| 15 | Shapiro-Wilk P-Value for Normality Test for TUV <sub>joint</sub> Data – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | Х |
| 16 | Shapiro-Wilk P-Value for Normality Test for TUV <sub>joint</sub> Data – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| 17 | Predictive Value of Planar Scans for SPECT/CT Per Joint and Reader (ITD Population) | Х | Х |
| 18 | Predictive Value of Planar Scans for SPECT/CT Per Joint and Reader (PP Population) | Х | |
| 19 | Number and Percentage of Subjects with TEAEs (Safety Population) | Х | Х |
| 20 | Summary of TEAEs (Safety Population) | Х | Х |
| 21 | Number and Percentage of Subjects with TESAEs (Safety Population) | Х | Х |
| 22 | Number and Percentage of Subjects With TEAEs by Severity Grade (Safety Population) | Х | Х |
| 23 | Number and Percentage of Subjects With TEAEs by Level of Relationship to Tc 99m Tilmanocept (Safety Population) | Х | Х |
| 24 | Number and Percentage of Subjects With TEAEs by Level of Relationship to Procedure (Safety Population) | Х | |

| Table<br>No. | Table Title | Included<br>in Final<br>Tables | Shown in<br>Appendix<br>B |
|---|---|---|---|
| 25 | Serum Chemistry Clinical Laboratory Parameters Summary Statistics by Arm (Safety Population) | X | X |
| 26 | Hematology Clinical Laboratory Parameters Summary Statistics by Arm (Safety Population) | X | |
| 27 | Urinalysis Clinical Laboratory Parameters Summary Statistics by Arm (Safety Population) | X | |
| 28 | Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | Х |
| 29 | Hematology Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | |
| 30 | Urinalysis Clinical Laboratory Parameters Shift Table by Arm (Safety Population) | Х | |
| 31 | Vital Signs Summary Statistics by Arm (Safety Population) | Χ | Х |

| Figure<br>No. | Figure Title | Included<br>in Final<br>Figures | Shown in<br>Appendix<br>B |
|---|---|---|---|
| Fig1 | Normal QQ plot for TUV <sub>joint</sub> Data – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | X |
| Fig2 | Normal QQ plot for TUV <sub>joint</sub> Data – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig3 | Scatter Plot of TUV <sub>joint</sub> Distribution of the Right Hand – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | Х |
| Fig4 | Scatter Plot of TUV <sub>joint</sub> Distribution of the Right Hand – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig5 | Scatter Plot of TUV <sub>joint</sub> Distribution of the Left Hand – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | Х |
| Fig6 | Scatter Plot of TUV <sub>joint</sub> Distribution of the Left Hand – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig7 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP1 by Age – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | Х |
| Fig8 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP1 by Age – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig9 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP2 by Age – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | |
| Fig10 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP2 by Age – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig11 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP3 by Age – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | |
| Fig12 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP3 by Age – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig13 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP4 by Age – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | |
| Fig14 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP4 by Age – All Arm 1 and 2 Healthy Control Subjects (PP Population) | Х | |
| Fig15 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP5 by Age – All Arm 1 and 2 Healthy Control Subjects (ITD Population) | Х | |

| Figure | | Included in Final | Shown in Appendix |
|---|---|---|---|
| No. | Figure Title | Figures | В |
| Fig16 | Scatter Plot of TUV <sub>joint</sub> Distribution for MCP5 by Age – All Arm 1 | Х | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig17 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP1 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig18 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP1 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig19 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP2 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig20 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP2 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig21 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP3 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig22 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP3 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig23 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP4 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig24 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP4 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig25 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP5 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig26 | Scatter Plot of TUV <sub>joint</sub> Distribution for PIP5 by Age – All Arm 1 | X | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig27 | Scatter Plot of TUV <sub>joint</sub> Distribution for Wrist by Age – All Arm 1 | Х | |
| | and 2 Healthy Control Subjects (ITD Population) | | |
| Fig28 | Scatter Plot of TUV <sub>joint</sub> Distribution for Wrist by Age – All Arm 1 | Х | |
| | and 2 Healthy Control Subjects (PP Population) | | |
| Fig29 | Scatter Plot of TUV <sub>joint</sub> Distribution by Sex – All Arm 1 and 2 | X | |
| | Healthy Control Subjects (ITD Population) | | |
| Fig30 | Scatter Plot of TUV <sub>joint</sub> Distribution by Sex – All Arm 1 and 2 | X | |
| | Healthy Control Subjects (PP Population) | | |
| Fig31 | Scatter Plot of TUV <sub>joint</sub> Distribution by BMI – All Arm 1 and 2 | X | |
| | Healthy Control Subjects (ITD Population) | | |
| Fig32 | Scatter Plot of TUV <sub>joint</sub> Distribution by BMI – All Arm 1 and 2 | Х | |
| | Healthy Control Subjects (PP Population) | | |
| Fig33 | Scatter Plot of Residuals by Age – All Arm 1 and 2 Healthy | X | X |
| | Control Subjects (ITD Population) | | |
| Fig34 | Scatter Plot of Residuals by Age – All Arm 1 and 2 Healthy | X | |
| | Control Subjects (PP Population) | | |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix<br>B |
|---|---|---|---|
| DL1 | Subject Disposition Data Listing | X | X |
| DL2 | Inclusion/Exclusion Data Listing | Х | Х |
| DL3 | Protocol Deviations Data Listing | Х | Х |
| DL4 | Demographics Data Listing | Х | Х |

| Listing<br>No. | Data Listing Title | Included<br>in Final<br>Listings | Shown in<br>Appendix<br>B |
|---|---|---|---|
| DL5 | Subjects Excluded from ITD Population Data Listing | X | X |
| DL6 | Subjects Excluded from PP Population Data Listing | X | X |
| DL7 | Subjects Excluded from Safety Population Data Listing | X | X |
| DL8 | Medical History Data Listing | X | Х |
| DL9 | Prior and Concomitant Medications Data Listing | X | Х |
| DL10 | Prior and Concomitant RA Medications Data Listing | Х | Х |
| DL11 | Adverse Events Data Listing | Х | Х |
| DL12 | Subject Laboratory Profiles – Hematology Data Listing | Х | Х |
| DL13 | Subject Laboratory Profiles – Serum Chemistry Data Listing | Х | |
| DL14 | Subject Laboratory Profiles – Urinalysis Data Listing | Х | |
| DL15 | Subject Laboratory Profiles – Rheumatology Panel Data Listing | Х | |
| DL16 | Physical Exam Data Listing | Х | Х |
| DL17 | ACR/EULAR 2010 Classification Data Listing | Х | Х |
| DL18 | DAS-28 by Joint Data Listing – Arm 2 RA Subjects | Х | Х |
| DL19 | DAS-28 by Subject Data Listing – Arm 2 RA Subjects | Х | Х |
| DL20 | Vital Signs Data Listing | Х | Х |
| DL21 | Study Drug Administration Data Listing | Х | Х |
| DL22 | Post-Injection Imaging Data Listing | Х | Х |
| DL23 | SPECT/CT Reader Results Data Listing – Hands and Wrists | Х | Х |
| DL24 | TUV Data Listing | Х | Х |

#### 8.0 References

Food & Drug Administration Center for Drug Evaluation and Research and Center for Biologics Evaluation and Research (September 1998). Guidance for Industry: ICH E9 Statistical Principles for Clinical Trials.

Forkman, J. (2009) Estimator and Tests for Common Coefficients of Variation in Normal Distributions. *Communications in Statistics: Theory and Methods*. 38:2, pp233-251.

# **Appendix A – Tables, Figures and Listing Specifications**

#### Orientation

Tables and figures will be displayed in landscape.

#### **Margins**

Margins will be 1 inch on all sides. Table and listing boundaries will not extend into the margins.

#### **Font**

Courier New, 8 point.

#### Headers

The table number will be on the first line of the title. The title area will contain the Sponsor name, the study number, and the name of the table. The title area will contain the page number (Page x of y) on the far right, 1 line above the name of the table.

#### **Footers**

- The first line will be a solid line.
- Next will be any footnotes regarding information displayed in the table.
- Below these footnotes will be displayed "STATKING Clinical Services (DD-MMM-YYYY)" on the far left.
- The last line will display the name of the SAS program that generated the table and (if applicable) the source data reference.

### **Table Disclaimer**

The format of the mock tables shown in the appendix of this SAP will be the format of the deliverable tables to the extent that Word document constructed tables can match production tables produced by SAS. This formatting includes the content and format of the header and footer areas of the tables. The Sponsor agrees to the format of the tables as shown in the appendix.

Further programming charges will be applicable for changes in the format of tables (including title statements, notes, data dependent footnotes, etc.) made after the approval of the SAP.

# **Missing Values**

All missing values will be displayed on the output tables/listings as blanks.

# **Display of Study Dates**

The date format to be used is dd-mmm-yyyy. Missing parts of dates are not shown (i.e., for a missing day value, the value displayed is in yyyy-mm format).

# Appendix B – Table Shells

Table 1. Subject Disposition by Study Arm Navidea Biopharmaceuticals - Study No. NAV3-35

| | | HC-1 | HC-2 | RA | Overall |
|---|---|---|---|---|---|
| | | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| Screen Failures | | | | | XX |
| Enrolled | | xxx | xxx | xxx | xxx |
| Completed | | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| Withdrawn | | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| Withdrawal Reason | Adverse Event | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Protocol Violation<br>Lost to Follow Up | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Withdrawal of Consent | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Sponsor Discretion | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Investigator Discretion | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Death | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |
| | Other | xx (xxx%) | xx (xxx%) | xx (xxx%) | xx (xxx%) |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) The denominator for all percentages in the table is the number of enrolled subjects in the respective arm and overall. STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Table 2. Demographics and Baseline Data Summary Statistics by Arm - Continuous Variables Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| Variable | Arma | Mean | Std Dev | n | Min | Max | Median |
|-----------------|------|------|---------|-----|-----|-----|--------|
| Age (years) | HC-1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA | XXX | XXX | XXX | XXX | XXX | XXX |
| Height (inches) | HC-1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA | XXX | XXX | XXX | XXX | XXX | XXX |
| Weight (pounds) | HC-1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA | XXX | XXX | XXX | XXX | XXX | XXX |
| BMI (kg/m^2) | HC-1 | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | XXX | XXX | XXX | XXX | XXX | XXX |
| | RA | XXX | XXX | XXX | XXX | XXX | XXX |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table 3. Demographics and Baseline Data Summary Statistics by Arm - Categorical Variables

Navidea Biopharmaceuticals - Study No. NAV3-35

Safety Population (N= xxx)

| | | | Arma | |
|---|---|---|---|---|
| | | HC-1 | HC -2 | RA |
| Variable | Category | (N= xxx) | (N= xxx) | (N= xxx) |
| Gender | Male | vvv (vvv%) | vvv (vvv%) | vvv (vvv%) |
| Gender | | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Female With Childbearing Potential | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Female With No Childbearing Potential | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Race | American Indian or Alaska Native | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Asian | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Black or African American | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Native Hawaiian or Other Pacific Islander | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | White | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Other | | | |
| Ethnicity | Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| 2 | Not Hispanic or Latino | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| II | Dialet Hended | /8 \ | | (° ) |
| Handedness | Right Handed | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Left Handed | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| | Ambidextrous | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table 4. Summary of Study Drug Administration by Arm
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N= xxx)

| | Arma | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|
| Tc 99m Dose (mCi) | HC-1 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | HC-2 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| Mass Dose (µg) | HC-1 | xxxx | XXXX | xx | xxxx | xxxx | xxxx |
| (r.g) | HC-2 | XXXX | xxxx | XX | XXXX | XXXX | XXXX |
| | RA | XXXX | xxxx | XX | XXXX | XXXX | XXXX |
| Total Volume of Tc 99m Tilmanocept Injected (mL) | HC-1 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | HC-2 | XXXX | XXXX | XX | XXXX | XXXX | XXXX |
| | RA | XXXX | XXXX | XX | XXXX | XXXX | XXXX |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 5. Summary of TUV<sub>joint</sub> on both Arms Per Reader, Joint, and View
Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

| Arma | Reader | View | Joint | Mean | Std Dev | n | Min | Max | Median |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | XXXXXXXXXXXXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | xxxxxxxxxxxxx | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| XXXX | XXXXXXXXXXXXXXX | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | xxxx.x | xxxx.x | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | xxxxxxxxxxxxx | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | xxxx.x | xxxx.x | XXXX.X |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | xxxx.x | xxxx.x | XXXX.X |
| | | xxxxxxxx | XX | XXXX.X | XXXX.X | XXX | XXXX.X | xxxx.x | xxxx.x |
| | | XXXXXXXX | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |

Table format is repeated for the PP population.

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 7. Summary of SUV on Arm 2 per Joint and Total of All Joints
Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

| Arm 2ª | Joint | Mean | Std Dev | n | Min | Max | Median |
|--------|--------------|--------|---------|-----|--------|--------|--------|
| HC-2 | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | Total of All | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | Joints | | | | | | |
| RA | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | XXXX.X |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | xxxx.x | XXXX.X |
| | XX | XXXX.X | XXXX.X | XXX | XXXX.X | XXXX.X | xxxx.x |
| | Total of All | XXXX.X | XXXX.X | xxx | XXXX.X | XXXX.X | xxxx.x |
| | Joints | | | | | | |

Table format is repeated for the PP population.

a HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Table 9. Normal Range of  $TUV_{joint}$  for the Three Blinded Readers in All Arm 1 and 2 Healthy Control Subjects

Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

| Joint | View | Reader | Number of<br>Joints | Mean | Standard<br>Deviation | Estimated<br>5 %tile | Estimated<br>95 %tile |
|---|---|---|---|---|---|---|---|
| xxxxxxxxxx | xx | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xx |
| | | xx | xxx | xxx.xx | xx.xx | xx.xxx | xx.xx |
| | | xx | xxx | xxx.xx | xx.xx | xx.xxx | xx.xx |
| | XX | xx | xxx | xxx.xx | XX.XXX | xx.xxx | xx.xxx |
| | | xx | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |
| | | XX | xxx | xxx.xx | xx.xxx | xx.xxx | xx.xxx |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

#### Table format is repeated for the PP population

Page x of y

Table 11. Correlation Between  $TUV_{joint}$  and Age and BMI - All Arm 1 and 2 Healthy Control Subjects Navidea Biopharmaceuticals - Study No. NAV3-35 ITD Population (N=xxx)

| Variable | TUV | P-value <sup>a</sup> |
|----------|--------|----------------------|
| AGE | xx.xxx | x.xxxx |
| BMI | xx.xxx | x.xxxx |

#### Table format is repeated for the PP population

<sup>&</sup>lt;sup>a</sup> P-value testing H0: Correlation Coefficient = 0 vs H1: Correlation Coefficient ≠ 0. STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas
Page x of y

Table 13. Frequency Counts and Percentage of Localization in SPECT/CT Imaging in RA Subjects
Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

#### Localized on SPECT/CT

| Joint | Reader | No | Yes | Total |
|-------------|--------|-------|-------|-------|
| XXXXXXXXXXX | XX | XXX | XXX | XXX |
| | | xx.x% | XX.X% | |
| | XX | XXX | xxx | XXX |
| | | XX.X% | XX.X% | |
| | xx | xxx | xxx | xxx |
| | | XX.X% | XX.X% | |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Table format is repeated for the PP population.

Page x of y

Table 15. Shapiro-Wilk P-Value for Normality Test for TUV<sub>joint</sub> Data - All Arm 1 and 2 Healthy Control Subjects

Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

Test for Normality

| Test | Statistic | P-Value |
|--------------|-----------|---------|
| Shapiro-Wilk | xxx | xxx |

STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

All Table format is repeated for the PP population

Page x of y

Table 17. Predictive Value of Planar Scans for SPECT/CT Per Joint and Reader
Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)

SPECT/CT (Standard of Truth)

| Reader | Joint | Planar Scans | Positive | Negative | Total | Uncertainty<br>Coefficients | Estimated<br>95 %tile |
|---|---|---|---|---|---|---|---|
| XX | XXX | TUVjoint > 95 (Positive) | XXX | XXX | XXX | XXX | XXX |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | XXX | XXX | | |
| | xxx | TUVjoint > 95 (Positive) | XXX | xxx | xxx | xxx | XXX |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | XXX | XXX | | |
| xx | xxx | TUVjoint > 95 (Positive) | XXX | XXX | xxx | XXX | XXX |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | XXX | XXX | | |
| | xxx | TUVjoint > 95 (Positive) | xxx | XXX | XXX | XXX | xxx |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | xxx | XXX | | |
| xx | xxx | TUVjoint > 95 (Positive) | xxx | XXX | xxx | xxx | XXX |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | xxx | XXX | | |
| | xxx | TUVjoint > 95 (Positive) | xxx | xxx | xxx | XXX | xxx |
| | | Negative | XXX | XXX | XXX | | |
| | | Total | XXX | XXX | XXX | | |

If there are no major protocol deviations, then analysis tables for the ITD and PP populations will contain identical results. STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

#### All Table format is repeated for the PP population

Page x of y

Table 19. Number and Percentage of Subjects with TEAEs
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N= xxx)

| Adverse Event Categoryb: | HC-1 | HC-2 | RA | Overall |
|---|---|---|---|---|
| Total Number of TEAEs | xxx | xxx | XXX | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Adverse events coded with MedDRA Coding Dictionary Version XXX

Page x of y

# Table 20. Summary of TEAEs Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| | | Arma | | |
|---|---|---|---|---|
| | HC-1 | HC-2 | RA | Overall |
| Subjects With at Least One TEAE | xxx | xxx | XXX | xxx |
| Maximum TEAE Severity Grade | | | | |
| Mild | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Moderate | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Severe | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Tc 99m tilmanocept | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Highest Relationship of TEAE to Study Procedure | | | | |
| Definitely Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably Not [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Possibly [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Probably [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Definitely [n(%)] | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 21. Number and Percentage of Subjects with TESAEs
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | | Arma | | |
|---|---|---|---|---|
| Adverse Event Categoryb: | HC-1 | HC-2 | RA | Overall |
| Total Number of TESAEs | xxx | xxx | xxx | xxx |
| Subjects with at Least One TESAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Adverse events coded with MedDRA Coding Dictionary Version XXX

Page x of y

Table 22. Number and Percentage of Subjects With TEAEs by Severity Grade
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

Part 1 of  $4 - HC-1^a$ 

| | Severity Grade | | |
|---|---|---|---|
| Adverse Event Categoryb: | Mild | Moderate | Severe |
| Total Number of TEAEs | xxx | xxx | xxx |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

STATKING Clinical Services (DD-MMM-YYYY)

Source Program: xxxxxxx.sas

Table format repeats for HA-2, RA (Parts 2 and 3) and overall (Part 4).

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Adverse events coded with MedDRA Coding Dictionary Version XXX

Page x of y

Table 23. Number and Percentage of Subjects With TEAEs by Level of Relationship to Tc 99m Tilmanocept

Navidea Biopharmaceuticals - Study No. NAV3-35

Safety Population (N=xxx)

Part 1 of 4 :  $HC-1^a$ 

Level of Relationship

| | Definitely | Probably | Possibly | Probably | Definitely |
|---|---|---|---|---|---|
| Adverse Event Categoryb: | Not | Not | Related | Related | Related |
| Total Number of TEAEs | XXX | XXX | XXX | XXX | XXX |
| Subjects with at Least One TEAE | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| System Organ Class 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 1 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| Preferred Term 2 | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Source Program: xxxxxxx.sas

Table format repeats for HC-2, RA (Parts 2 and 3) and overall (Part 4). Full Table (all parts) repeats for Table 24.

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Adverse events coded with MedDRA Coding Dictionary Version XXX STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 25. Serum Chemistry Clinical Laboratory Parameters Summary Statistics by Arm
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | | | | | Std | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter(units) | $\operatorname{Arm}^{\operatorname{a}}$ | Visit | Data Type <sup>b</sup> | Mean | Dev | n | Min | Max | Median |
| xxxxxxxx (xxx) | HC-1 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Visit 2) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Visit 2) | RAW | | | | | | |
| | | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |
| | RA | Screening (Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Visit 2) | RAW | | | | | | |
| | | | CFB | XXX | XXX | xxx | XXX | XXX | XXX |
| xxxxxxx (xxx) | HC-1 | Screening (Baseline) | RAW | xxx | xxx | xxx | xxx | XXX | xxx |
| | | Day 0 (Visit 2) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | Screening (Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Visit 2) | RAW | | | | | | |
| | | | CFB | xxx | XXX | XXX | XXX | XXX | XXX |
| | RA | Screening (Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 (Visit 2) | RAW | | | | | | |
| | | | CFB | xxx | XXX | XXX | XXX | XXX | xxx |

Source Program: xxxxxxx.sas

Table format repeats for Tables 26 and 27.

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value) STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Table 28. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

Part 1 of 3: HC-1a

### Baseline Result/ Post-Injection Result

| Panel/Parameter (units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx(xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table format is repeated for Tables 29 (Hematology) and 30 (Urinalysis)

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 28. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

Part 2 of 3: HC-2a

## Baseline Result/ Post-Injection Result

| Panel/Parameter (units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx)<br>xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table format is repeated for Tables 29 (Hematology) and 30 (Urinalysis)

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 28. Serum Chemistry Clinical Laboratory Parameters Shift Table by Arm
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

Part 3 of 3: RAa

### Baseline Result/ Post-Injection Result

| Panel/Parameter (Units) | Low/<br>Low | Low/<br>Normal | Low/<br>High | Normal/<br>Low | Normal/<br>Normal | Normal/<br>High | High/<br>Low | High/<br>Normal | High/<br>High |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | XXX (XXX°) | XXX (XXX%) | xxx (xxx%) | xxx (xxx%) | XXX (XXX°) | XXX (XXX°) | XXX (XXX°) | XXX (XXX <sup>5</sup> ) | XXX (XXX%) |
| xxxxxxx/ | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |
| xxxxxxxx (xxx) | | | | | | | | | |
| xxxxxxx/<br>xxxxxxxx (xxx) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) | xxx (xxx%) |

Table format is repeated for Tables 29 (Hematology) and 30 (Urinalysis)

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Table 31. Vital Signs Summary Statistics by Arm Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| Vital Sign | | | Data | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Parameter (units) | ${\tt Arm^a}$ | Visit | Type <sup>b</sup> | Mean | Std Dev | n | Min | Max | Median |
| xxxxxxxxx (xxx) | HC-1 | Screening | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | Screening | RAW | xxx | XXX | xxx | xxx | xxx | xxx |
| | | | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | XXX |
| | HC-2 | Day 0 Pre-Injection(Baseline) | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | Day 0 Post-Injection | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | XXX | xxx |
| | RA | Screening | RAW | xxx | XXX | xxx | xxx | xxx | xxx |
| | | | RAW | xxx | XXX | XXX | XXX | XXX | XXX |
| | | | CFB | XXX | XXX | XXX | XXX | xxx | XXX |
| | RA | Day 0 Pre-Injection(Baseline) | RAW | XXX | XXX | XXX | XXX | xxx | XXX |
| | | Day 0 Post-Injection | RAW | XXX | XXX | XXX | XXX | xxx | XXX |
| | | | CFB | xxx | xxx | xxx | xxx | xxx | XXX |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b RAW = data recorded in database; CFB = change from baseline= (parameter value at the current time point)-(Baseline parameter value). STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Figure 1. Normal QQ plot for  $TUV_{joint}$  Data - All Arm 1 and 2 Healthy Control Subjects Navidea Biopharmaceuticals - Study No. NAV3-35 ITD Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format is repeated for the PP population.

Page x of y

Figure 3. Scatter Plot of  $TUV_{joint}$  Distribution of the Right Hand - All Arm 1 and 2 Healthy Control Subjects Navidea Biopharmaceuticals - Study No. NAV3-35 ITD Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format is repeated for the PP population.

Page x of y

Figure 5. Scatter Plot of TUVjoint Distribution of the Left Hand - All Arm 1 and 2 Healthy Control Subjects

Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format is repeated for the PP population.

Page x of y

Figure 7. Scatter Plot of TUV<sub>joint</sub> Distribution for MCP1 by Age - All Arm 1 and 2 Healthy Control Subjects

Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format is repeated per joint and again for the PP population per joint. Repeat for Sex and BMI.

Page x of y

Figure 33. Scatter Plot of Residuals by Age - All Arm 1 and 2 Healthy Control Subjects

Navidea Biopharmaceuticals - Study No. NAV3-35

ITD Population (N=xxx)



STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Figure format is repeated the PP Population.

Page x of y

Data Listing 1. Subject Disposition Data Listing Navidea Biopharmaceuticals - Study No. NAV3-35

| | Subject | | | |
|---|---|---|---|---|
| Arma | No. | Disposition Status | Withdrawal | Withdrawal Reason |
| XXXXXX | xxxx | xxxxxxxxxxxxxxxxx | xxxxxxxx | ****** |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | XXXXXXXXXXXXXXXXXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx |

oodioo iiogiam. mmmmiiiodo

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 2. Inclusion/Exclusion Data Listing Navidea Biopharmaceuticals - Study No. NAV3-35

| Arm <sup>a</sup> | Subject<br>No. | Did Subject<br>Meet All<br>Eligibility<br>Criteria? | Criterion Category | Criterion | Was a<br>Waiver<br>Granted? | Is Subject a<br>Screen<br>Failure? |
|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXXXX | XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXXXX | XXXX | XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX | XXXX | XXXX |
| XXXXXX | XXXX | xxxx | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx | XXXX | xxxx |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 3. Protocol Deviations Data Listing Navidea Biopharmaceuticals - Study No. NAV3-35

| Arm <sup>a</sup> | Subject<br>No. | Date of<br>Deviation | Deviation Description | Deviation Category<br>(Major/Minor) |
|---|---|---|---|---|
| XXXXXX | XXXX | XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxx |
| XXXXXX | XXXX | XXXXXX | xxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXX |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 4. Demographics Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=135)

| Armª | Subject<br>No. | Informed<br>Consent<br>Date/Time | Date<br>of<br>Birth | Height<br>(inches) | Weight<br>(pounds) | Age<br>(yrs) | Gender | Race | Ethnicity | Handedness | WOCBP? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | _ |
| XXXXXX | XXXX | XXXXXX | XXXXXX | XXX | XXX | XXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 5. Subjects Excluded from ITD Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|-------------------------|
| • | | |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxxx.sas

Page x of y

Data Listing 6. Subjects Excluded from PP Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|--------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxxx.sas

Page x of y

Data Listing 7. Subjects Excluded from Safety Population Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
All Enrolled Subjects (N=xxx)

| Arma | Subject No. | Reason for Exclusion |
|--------|-------------|--------------------------|
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxxx.sas

Page x of y

Data Listing 8. Medical History Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | | MedDRA System Organ Classb/ | | | |
|---|---|---|---|---|---|
| | Subject | MedDRA Preferred Term/ | Resolution/Stop | | |
| Arma | No. | CRF Verbatim Term | Start Date | Date | Ongoing? |
| XXXXXX | XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXX |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Medical history terms coded with MedDRA Coding Dictionary Version xxx. STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 9. Prior and Concomitant Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

Drug Preferred Termb/

| | | verbatim/ | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject ATC Level 1 Text/ | | | | Start | Stop | | |
| Arma | No. | ATC Level 4 Text | Indication | Frequency | Date | Date | Route | Ongoing? |
| XXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| XXXXXX | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 10. Prior and Concomitant RA Medications Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

 ${\tt Drug\ Preferred\ Term^b/}$ 

| | | Verbatim/ | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Subject | ATC Level 1 Text/ | | | Start | Stop | | |
| Arma | No. | ATC Level 4 Text | Indication | Frequency | Date | Date | Route | Ongoing? |
| | | | | | | | | _ |
| XXXXXX | XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| XXXXXX | XXXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | XXXXX | XXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
| | | xxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Medications coded with WHO Coding Dictionary xxxxxxxxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 11. Adverse Events Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | | Start | | | MedDRA System Organ | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Date and | Start Date | | Class <sup>b</sup> / | | Relation to | | |
| | | Time/ | and Time of | | MedDRA Preferred | | Tc-99m | | |
| | Subject | End Date | tilmanocept | Treatment | Term/ | | tilmanocept/ | | |
| ${\tt Arm^a}$ | No. | and Time | Injection | Emergent? | CRF Verbatim Term | Severity | Procedure | Serious? | Outcome |
| XXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxxx | XXXXXXXX | xxxxxxxx/ | XXX | XXXXXXXX |
| | | xxxxxxx/ | | | xxxxxxxxxxxxxx | | XXXXXXX | | |
| | | XXXXXXX | | | xxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | | | | | | |
| XXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXX | xxxxxxxxxxxxx | XXXXXXX | xxxxxxxx/ | XXX | XXXXXXX |
| | | xxxxxxx/ | XXXXXXX | | xxxxxxxxxxxxxxx | | XXXXXXX | | |
| | | XXXXXXX | | | xxxxxxxxxxxxxxx | | | | |
| | | XXXXXXX | | | | | | | |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Adverse events coded with MedDRA Coding Dictionary Version xxx STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 12. Subject Laboratory Profiles - Hematology Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | | | | | | | Norma | | |
|---|---|---|---|---|---|---|---|---|---|
| _ | Arm <sup>a</sup> | Subject<br>No. | Visit | Sample Date<br>and Time | Lab Parameter (Units) | Result | Lab Low | Lab High | Clin. Sig? |
| | XXXXXX | XXXX | XXXXXXX | xxxxxxxx / xx:xx | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | XXX | XXX | XXX | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | xxx | xxx | xxx | XXX |
| | | | | | xxxxxxxxxxxx (xxx) | XXX | XXX | xxx | XXX |

Table format is repeated for Serum Chemistry, Urinalysis, and Rheumatology Panel Listings (Listings 13, 14, 15).

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 16. Physical Exam Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | Subject | | Date | | | |
|---|---|---|---|---|---|---|
| ${\tt Arm^a}$ | No. | Visit | Conducted | Body System | Result | Abnormality |
| XXXXXX | XXXX | XXXXXXX | XXXXXXX | General Appearance | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Skin | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Eyes, Ears, Nose, Throat | XXXXXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Head and Neck | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lungs | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Heart | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Abdomen | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Lymph Nodes | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Musculoskeletal | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Nervous System | xxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | | | | Other: XXXXXX | xxxxxxxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 17. ACR/EULAR 2010 Classification Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

ACR/EULAR 2010

| Arma | Subject | Visit | Date | Joint<br>Involvement | Serology | Acute-<br>Phase<br>Reactants | Duration<br>of<br>Symptoms | Total Score |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxx | xxxxxxx | xxx | XXX | XXX | XXX | xxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxx | xxx | xxx | xxx | xxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

Data Listing 18. DAS-28 by Joint Data Listing - Arm 2 RAª Subjects
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

#### DAS28 Joint Classification

| Subject | | | | Result | Result |
|---------|---------|---------|----------|--------------|-------------|
| No. | Visit | Date | Joint | (Right Body) | (Left Body) |
| XXXX | XXXXXXX | XXXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| XXXX | XXXXXX | XXXXXX | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |
| | | | XXXXXXXX | XXX | XXX |

<sup>&</sup>lt;sup>a</sup> RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 19. DAS-28 by Subject Data Listing - Arm 2 RA $^{\rm a}$  Subjects Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| | | | | | DAS28 | | |
|---|---|---|---|---|---|---|---|
| | | • | | | Patient | Erythrocyte | |
| | | | Tender | Swollen | VAS | Sedimentation | |
| Subject | | | Joint | Joint | Global | Rate (ESR; | DAS28 |
| No. | Visit | Date | Count | Count | (mm) | mm/hr) | Score |
| XXXX | xxxxxxx | xxxxxx | XXX | xxx | xxx | xxx | xxx |
| xxxx | xxxxxxx | xxxxxxx | xxx | xxx | xxx | xxx | xxx |

a RA = rheumatoid arthritis (stable treatment regimen; Arm 2)
STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 20. Vital Signs Data Listing Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| | | | | | | Systolic<br>Blood | Diastolic<br>Blood | Heart | |
|---|---|---|---|---|---|---|---|---|---|
| | Subject | | | | Temp. | Pressure | Pressure | Rate | Respirations |
| Arma | No. | Visit | Date | Time | (°F) | (mmHg) | (mmHg) | (bpm) | per Minute |
| xxxxxx | xxxx | xxxxxxx | xxxxxxx | xxxxx | xxx | xxx | xxx | xxx | xxx |
| | | | | xxxxx | XXX | XXX | xxx<br>xxx | XXX<br>XXX | xxx<br>xxx |
| xxxxxx | xxxx | xxxxxx | xxxxxxx | xxxxx | xxx | xxx | xxx | xxx | xxx |
| | | | | XXXXX | xxx | xxx<br>xxx | xxx<br>xxx | xxx | xxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY)

Page x of y

Data Listing 21. Study Drug Administration Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| Arm <sup>a</sup> | Subject<br>No. | Date/<br>Time of<br>Injection | Anatomic<br>Location<br>of<br>Injection | Pre-Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Post-<br>Injection<br>Radioactivity<br>(mCi)/Time of<br>Measurement | Calculated Amount of Administered Radioactivity (mCi) | Source<br>Recorded<br>Administered<br>Radioactivity<br>(mCi) | Calculated<br>Mass Dose<br>(µg) | Volume<br>Injected<br>(mL) | Lot<br>Number |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx | xxx |
| xxxxxx | xxxx | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | xxx | xxx |
| | | xxxxxxxx/<br>xxxx | xxxxxxx | xxx/<br>xxxx | xxx/<br>xxxx | xxx | xxx | xxx | XXX | xxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)STATKING Clinical Services (DD-MMM-YYYY)
Source Program: xxxxxxx.sas

Page x of y

Data Listing 22. Post-Injection Imaging Data Listing
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| | Arm <sup>a,b</sup> | Subject<br>No. | Visit | Date of<br>Imaging | Start Time<br>of Planar<br>Imaging | End Time<br>of Planar<br>Imaging | Start Time<br>of SPECT/CT<br>Imaging | End Time<br>of SPECT/CT<br>Imaging |
|---|---|---|---|---|---|---|---|---|
| - | xxxxxx | xxxx | xxxxxxx | xxxxxx | xx:xx | xx:xx | xx:xx | xx:xx |
| | xxxxxx | xxxx | xxxxxxx | xxxxxx | xx:xx | xx:xx | xx:xx | xx:xx |

STATKING Clinical Services (DD-MMM-YYYY)

a HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

 $<sup>^{\</sup>rm b}$  SPECT/CT imaging performed only in study Arm 2 - RA

Page x of y

Data Listing 23. SPECT/CT Reader Results Data Listing - Hands and Wrists
Navidea Biopharmaceuticals - Study No. NAV3-35
Safety Population (N=xxx)

| Arma | Subject<br>No. | Post-Injection<br>Imaging Time Point | Joint | SPECT/CT<br>Localization? |
|---|---|---|---|---|
| xxxxxx | xxxx | xxxxxx | xxxxxxxxxx | xxxx |
| xxxxxx | xxxx | xxxxxx | XXXXXXXXXXX<br>XXXXXXXXXXX | xxxx |

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2) STATKING Clinical Services (DD-MMM-YYYY) Source Program: xxxxxxx.sas

Page x of y

# Data Listing 24. TUV Data Listing Navidea Biopharmaceuticals - Study No. NAV3-35 Safety Population (N=xxx)

| | Subject | | | Region of | |
|---|---|---|---|---|---|
| $\mathtt{Arm}^\mathtt{a}$ | No. | Visit | Date/Time | Interestb | TUV |
| xxxxxx | xxxx | xxxxxx | xxxxxxxxxxx | xxxxx | xxxxx |
| xxxxxx | xxxx | xxxxxxx | xxxxxxxxxxxx | XXXXXX | xxxxx |

STATKING Clinical Services (DD-MMM-YYYY)

<sup>&</sup>lt;sup>a</sup> HC-1 = healthy control-Arm 1, HC-2 = healthy control-Arm 2, RA = rheumatoid arthritis (stable treatment regimen; Arm 2)

b Region of Interest is joint for all arms, and joint or Global for the Arm 2 - RA.